CLINICAL TRIAL: NCT01798290
Title: Impact of an Educational Program 'Narrative Medicine (Workshop Reading Diaries) ' Dedicated to Medical Students. A Randomized Controlled Trial.
Brief Title: Impact of Narrative Medicine (Workshop Reading Diaries)
Acronym: INAMEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RAV002 INAMEDI
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2012-11

CONDITIONS: Empathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral: narrative medicine: reading workshop (Experimental): Students allocated to the active comparator arm will follow 5 sessions in Class-led instruction of reading patients' diaries or nurses'diaries. They will be divided into eight subgroups of 12 students. The first and fifth sessions will be presential, and 2nd 3rd and 4th sessions will be homework to do on internet.
  Interventions: Behavioral: narrative medicine: reading workshop
- Behavioral: critical reading (Active Comparator): Students allocated to the active comparator arm will follow 5 sessions in Class-led instruction of reading literature. They will be divided into eight subgroups of 12 students. The first and fifth sessions will be presential, and 2nd 3rd and 4th sessions will be homework to do on internet.
  Interventions: Behavioral: critical reading

INTERVENTIONS:
Behavioral: narrative medicine: reading workshop
  Arms: Behavioral: narrative medicine: reading workshop
Behavioral: critical reading
  Arms: Behavioral: critical reading

SUMMARY:
Objective: The aim of this study is to assess the impact of an educational program of Narrative Medicine "workshop reading diaries" dedicated to medical students on their empathy.

Design: Randomized Controlled Trial in 2 arms. Participants: Medical students (4th years) of the University Paris Descartes. Methods: participants will be randomized in 2 groups. The allocation of participants will be done by a computerized randomization list, the sequence will be created by an independent statistician. Participants will be blinded of the study hypothesis. Allocation concealment will be provided because only the statistician will have access to the randomization list.

A program of Narrative Medicine with lesson in small group of "workshop reading patients' diaries " vs "workshop reading literature".

Outcome: The primary endpoint will be a first measure of the empathy of the medical students. The secondary endpoints will be a second measure of the empathy of the medical student; satisfaction of the student relative to the educational program .

Potential interests: We believe that the workshop "reading patients' diaries" can develop the thinking of the student with respect to his behavior with the patient, and so the relation between student and patient.

Sample size expected: 200 participants.

ELIGIBILITY:
Inclusion Criteria:

* All students in the fourth year of medical

Exclusion Criteria:

* refuse to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The Jefferson Scale of Physician Empathy | 5 months after randomization (i.e. 1 month after the end of the intervention)
  self-administered questionnaire consisting of 20 items scored by a Likert-type scale (strongly agree = 7, strongly disagree = 1): 10 items are rated positively, others 10 items are rated negatively. The total score ranges from 20 to 140.

SECONDARY OUTCOMES:
The Interpersonal Reactivity Index | 5 months after randomization (i.e. 1 month after the end of the intervention)
  self-administered questionnaire with 4 subscales (Perspective Taking, Empathic Concern, Fantasy, Personal Distress) each containing seven items (a total of 28 items). The items are scored by a Likert scale (0 = Does not describe me well to 4 = Describes me very well).
students' satisfaction | 4 months after randomization (i.e. 1 month after the end of the intervention)
  measure on a numeric scale from 0 (without interest) to 10 (very interesting)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'épidémiologie clinique, Hôtel Dieu, Paris, France